CLINICAL TRIAL: NCT03044379
Title: A Randomized, Double Blind, Placebo-Controlled, Phase 1 Safety and Pharmacokinetic Study of Dapivirine Gel (0.05%) Administered Rectally to HIV-1 Seronegative Adults
Brief Title: Dapivirine Gel Rectal Safety and PK Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Current program is on hold, not for safety reason
Sponsor: International Partnership for Microbicides, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MTN-026/ IPM 038
Record Dates: First submitted 2016-09-06; First posted 2017-02-07 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-10

CONDITIONS: HIV 1 Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapivirine Gel (Active Comparator): Participants will be randomized to receive a single dose of dapivirine gel rectally, followed by 7 daily doses of the same product to be administered under direct observation in the clinic.
  Interventions: Drug: Dapivirine gel (0.05%)
- Placebo Gel HEC (Placebo Comparator): Participants will be randomized to receive the universal HEC placebo gel rectally, followed by 7 daily doses of the same product to be administered under direct observation in the clinic.
  Interventions: Other: Universal HEC placebo gel

INTERVENTIONS:
Drug: Dapivirine gel (0.05%) — MTN-026/IPM 038 will use the HTI pre-filled applicator, the same applicator that has been utilized in other rectal studies.
  Arms: Dapivirine Gel
Other: Universal HEC placebo gel
  Arms: Placebo Gel HEC

SUMMARY:
Dapivirine Gel Rectal Safety and PK Study

DETAILED DESCRIPTION:
A Randomized, Double Blind, Placebo-Controlled Phase 1 Safety and Pharmacokinetic Study of Dapivirine Gel (0.05%) Administered Rectally to HIV-1 Seronegative Adults

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 45 years (inclusive), verified per site SOP
* Able and willing to provide written informed consent
* HIV-1/2 uninfected at Screening and Enrollment, per applicable algorithm in Appendix II and willing to receive HIV test results
* Able and willing to provide adequate locator information, as defined in site SOP
* Available to return for all study visits and willing to comply with study participation requirements
* In general good health at Screening and Enrollment, as determined by the site IoR or designee
* Per participant report, a history of consensual RAI at least once in the past calendar year
* Willing to not take part in other research studies involving drugs, medical devices, genital products, or vaccines for the duration of study participation, including the time between Screening and Enrollment

Exclusion Criteria: At Screening:

* Hemoglobin Grade 1 or higher*
* Platelet count Grade 1 or higher*
* White blood count Grade 2 or higher*
* Serum creatinine 1.3 the site laboratory upper limit of normal (ULN)
* International normalized ratio (INR) 1.5 the site laboratory ULN
* Aspartate aminotransferase (AST) or alanine transaminase (ALT) Grade 1 or higher*
* Positive for hepatitis C antibody
* Positive for hepatitis B surface antigen
* History of inflammatory bowel disease by participant report

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09-29 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Safety To characterize the systemic and compartmental pharmacokinetics of dapivirine gel following rectal application. | 9-12 months
  To evaluate the safety of dapivirine gel formulation when applied rectally.

SECONDARY OUTCOMES:
Acceptability | 9-12 months
  To identify product attributes considered likely to challenge and facilitate future sustained use of rectally applied dapivirine gel.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No